CLINICAL TRIAL: NCT05997433
Title: Efficacy of 7-day Versus 14-day Bismuth Quadruple Therapy for the Eradication of Helicobacter Pylori : A Multicenter Randomized Non-Inferiority Trial
Brief Title: Efficacy of 7-day Versus 14-day Bismuth Quadruple Therapy for the Eradication of Helicobacter Pylori（SHARE2302)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Collaborators: Zibo Maternal and Child Health Hospital (Unknown); Zaozhuang Municipal Hospital (Other); Binzhou Maternal and Child Health Hospital (Unknown); Jinxiang County People's Hospital (Unknown); Linyi Yizhou Hospital (Unknown); Yantai Penglai Traditional Chinese Medicine Hospital (Unknown); Shandong University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Yanqing Li, Dr, Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHARE2302
Record Dates: First submitted 2023-08-11; First posted 2023-08-18 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Helicobacter Pylori Infection
MeSH Terms: interventions — Amoxicillin; Tetracycline; Bismuth; tegoprazan

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 7 days (Experimental): Amoxicillin 1000mg bid+ Tetracycline 500mg qid+ Bismuth + Tegoprazan 50mg bid
  Interventions: Procedure: 7days bismuth quadruple
- 14 days (Active Comparator): Amoxicillin 1000mg bid+ Tetracycline 500mg qid+ Bismuth + Tegoprazan 50mg bid
  Interventions: Procedure: 14 days bismuth quadruple

INTERVENTIONS:
Procedure: 7days bismuth quadruple — Amoxicillin 1000mg bid+ Tetracycline 500mg qid+ Bismuth + Tegoprazan 50mg bid*7days
  Other Names: Amoxicillin; Tetracycline; Bismuth; Tegoprazan
  Arms: 7 days
Procedure: 14 days bismuth quadruple — Amoxicillin 1000mg bid+ Tetracycline 500mg qid+ Bismuth + Tegoprazan 50mg bid*14days
  Other Names: Amoxicillin; Tetracycline; Bismuth; Tegoprazan
  Arms: 14 days

SUMMARY:
Helicobacter pylori (H. pylori) infection is a common global infectious disease of the gastrointestinal tract. Helicobacter pylori eradication can effectively prevent the development of gastric cancer.The researchers collect H.pylori-positive patients who need native therapy. The subjects were randomized to receive7 days and 14 days of bismuth quadruple eradication therapy. 6-8 weeks after treatment, the subjects will re-take the 13C-urea breath test. Calculate the eradication rates, adverse reaction rates and patient compliance of each group.

DETAILED DESCRIPTION:
Related studies have shown that 7-day bismuth quadruple therapy is not inferior to 14-day bismuth quadruple therapy in the eradication of clarithromycin-resistant H. pylori.The results of the current study conducted by our team on the eradication of H. pylori in 10-day versus 14-day courses of bismuth quadruple therapy showed that the 10-days (92.09%) was not inferior to the 14-days(92.38%), but the incidence of adverse effects was significantly lower in the 10-day courses than in the 14-days(30.62%). If it can be demonstrated that the eradication rate of the 7-day course of bismuth quadruplex is close to that of the 14-days, then the 7-day course may be chosen.

The researchers collect H.pylori-positive patients who need native therapy. If the subject meets the selection criteria but not the exclusion criteria, and signs an informed consent form, the researchers randomized the subjects in groups: subjects received 7days or 14days bismuth quadruple eradication therapy. The medication of groups are as follows. 6-8 weeks after the eradication treatment, the subjects will review the 13C-urea breath test, and the researcher records the results.

After all subjects were tested, the eradication rates, adverse reaction rates and patient compliance of each group were calculated.

According to therapy, it is randomized into a 7days treatment group and a 14 days treatment group. The two groups of bismuth quadruple regimens are the same, as follows:

7days group: Amoxicillin 1000mg bid+ Tetracycline 500mg qid+ Bismuth + Tegoprazan 50mg bid 14days group: Amoxicillin 1000mg bid+ Tetracycline 500mg qid+ Bismuth + Tegoprazan 50mg bid

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18-70.
2. Without active hepatitis.
3. Helicobacter pylori infection (either positive for rapid urease test, C13/C14 urea breath test).
4. Patients who have not previously received helicobacter pylori eradication therapy.

Exclusion Criteria:

1. Patients with serious underlying diseases, such as liver insufficiency (Aspartate aminotransferase or alanine aminotransferase greater than the normal value), renal insufficiency (Cr≥2.0mg/dL or glomerular filtration rate <50 ml/min), immunosuppression, malignant tumors, Coronary heart disease or coronary artery stenosis ≥75%.
2. Patients who are pregnant or lactating or unwilling to take contraceptive measures during the trial.
3. Patients with active gastrointestinal bleeding.
4. Patients with a history of upper gastrointestinal surgery.
5. Patients allergic to treatment drugs.
6. Patients with medication history of bismuth agents, antibiotics, proton pump inhibitor and other drugs within 4 weeks.
7. Patients with other behaviors that may increase the risk of illness, such as alcohol and drug abuse.
8. Patients who are unwilling or incapable to provide informed consents.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Estimated)
Dates: Start 2023-09-02 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Eradication rate | Immediately after follow-up check
  Both intention to treat (ITT) and per-protocol (PP) analyses will be used for the assessment of the eradication rates of Helicobacter pylori infections in two groups. The ITT analysis includes all randomly assigned patients who take at least one dose of the study medications. The PP analysis is limited to patients who take over 90% of the study medications and complete follow-up.

SECONDARY OUTCOMES:
Rate of adverse reactions | Immediately after follow-up check
  Rate of adverse reactions
Patient compliance | Immediately after follow-up check
  Good compliance is defined as the actual dosage is within the range of 90%-100% of the dosage that should be taken.

CONTACTS AND LOCATIONS:
Overall Officials: Yanqing Li, Ph.D, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China

REFERENCES:
- [Result] Hooi JKY, Lai WY, Ng WK, Suen MMY, Underwood FE, Tanyingoh D, Malfertheiner P, Graham DY, Wong VWS, Wu JCY, Chan FKL, Sung JJY, Kaplan GG, Ng SC. Global Prevalence of Helicobacter pylori Infection: Systematic Review and Meta-Analysis. Gastroenterology. 2017 Aug;153(2):420-429. doi: 10.1053/j.gastro.2017.04.022. Epub 2017 Apr 27. PMID 28456631
- [Result] Malfertheiner P, Megraud F, O'Morain C, Bazzoli F, El-Omar E, Graham D, Hunt R, Rokkas T, Vakil N, Kuipers EJ. Current concepts in the management of Helicobacter pylori infection: the Maastricht III Consensus Report. Gut. 2007 Jun;56(6):772-81. doi: 10.1136/gut.2006.101634. Epub 2006 Dec 14. PMID 17170018
- [Result] Cho JH, Jin SY. Current guidelines for Helicobacter pylori treatment in East Asia 2022: Differences among China, Japan, and South Korea. World J Clin Cases. 2022 Jul 6;10(19):6349-6359. doi: 10.12998/wjcc.v10.i19.6349. PMID 35979311
- [Result] Zhou XZ, Lyu NH, Zhu HY, Cai QC, Kong XY, Xie P, Zhou LY, Ding SZ, Li ZS, Du YQ; National Clinical Research Center for Digestive Diseases (Shanghai), Gastrointestinal Early Cancer Prevention & Treatment Alliance of China (GECA), Helicobacter pylori Study Group of Chinese Society of Gastroenterology and Chinese Alliance for Helicobacter pylori Study.. Large-scale, national, family-based epidemiological study on Helicobacter pylori infection in China: the time to change practice for related disease prevention. Gut. 2023 May;72(5):855-869. doi: 10.1136/gutjnl-2022-328965. Epub 2023 Jan 23. PMID 36690433
- [Result] Ding SZ, Du YQ, Lu H, Wang WH, Cheng H, Chen SY, Chen MH, Chen WC, Chen Y, Fang JY, Gao HJ, Guo MZ, Han Y, Hou XH, Hu FL, Jiang B, Jiang HX, Lan CH, Li JN, Li Y, Li YQ, Liu J, Li YM, Lyu B, Lu YY, Miao YL, Nie YZ, Qian JM, Sheng JQ, Tang CW, Wang F, Wang HH, Wang JB, Wang JT, Wang JP, Wang XH, Wu KC, Xia XZ, Xie WF, Xie Y, Xu JM, Yang CQ, Yang GB, Yuan Y, Zeng ZR, Zhang BY, Zhang GY, Zhang GX, Zhang JZ, Zhang ZY, Zheng PY, Zhu Y, Zuo XL, Zhou LY, Lyu NH, Yang YS, Li ZS; National Clinical Research Center for Digestive Diseases (Shanghai), Gastrointestinal Early Cancer Prevention & Treatment Alliance of China (GECA), Helicobacter pylori Study Group of Chinese Society of Gastroenterology, and Chinese Alliance for Helicobacter pylori Study. Chinese Consensus Report on Family-Based Helicobacter pylori Infection Control and Management (2021 Edition). Gut. 2022 Feb;71(2):238-253. doi: 10.1136/gutjnl-2021-325630. Epub 2021 Nov 26. PMID 34836916
- [Result] Liou JM, Malfertheiner P, Lee YC, Sheu BS, Sugano K, Cheng HC, Yeoh KG, Hsu PI, Goh KL, Mahachai V, Gotoda T, Chang WL, Chen MJ, Chiang TH, Chen CC, Wu CY, Leow AH, Wu JY, Wu DC, Hong TC, Lu H, Yamaoka Y, Megraud F, Chan FKL, Sung JJ, Lin JT, Graham DY, Wu MS, El-Omar EM; Asian Pacific Alliance on Helicobacter and Microbiota (APAHAM). Screening and eradication of Helicobacter pylori for gastric cancer prevention: the Taipei global consensus. Gut. 2020 Dec;69(12):2093-2112. doi: 10.1136/gutjnl-2020-322368. Epub 2020 Oct 1. PMID 33004546
- [Result] Moon SG, Lim CH, Kang HJ, Choi A, Kim S, Oh JH. Seven Days of Bismuth-Based Quadruple Therapy Is as Effective for the First-Line Treatment of Clarithromycin-Resistant Confirmed Helicobacter pylori Infection as 14 Days of Bismuth-Based Quadruple Therapy. J Clin Med. 2022 Jul 30;11(15):4440. doi: 10.3390/jcm11154440. PMID 35956057
- [Result] Qiao C, Li Y, Liu J, Ji C, Qu J, Hu J, Ji R, Wan M, Lin B, Lin M, Qi Q, Zuo X, Li Y. Clarithromycin versus furazolidone for naive Helicobacter pylori infected patients in a high clarithromycin resistance area. J Gastroenterol Hepatol. 2021 Sep;36(9):2383-2388. doi: 10.1111/jgh.15468. Epub 2021 Mar 10. PMID 33691344
- [Derived] Nan XP, Zhao HY, Guo LN, Zheng RQ, Wang XL, Wang YF, Su YH, Geng WR, Liu XL, Xu HM, Zhou KL, Guo YT, Cao JH, Han ZX, Kong QZ, Zuo XL, Li YQ, Li YY. Seven-Day Versus 14-Day Tegoprazan and Tetracycline-Containing Quadruple Therapy for First-Line Eradication of Helicobacter pylori Infection: A Randomized, Open-Label, Noninferiority Trial. Helicobacter. 2025 Mar-Apr;30(2):e70036. doi: 10.1111/hel.70036. PMID 40272011